CLINICAL TRIAL: NCT06311695
Title: The Role of Contrast-Enhanced Spectral Mammography (CESM) in the Diagnostic Process of Breast Cancer
Brief Title: Contrast-Enhanced Spectral Mammography (CESM)
Acronym: CESM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO 960
Record Dates: First submitted 2022-11-21; First posted 2024-03-15 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: mammography; enhancement; Contrast Enhanced Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contrast Enhanced Mammography (Experimental): Patients underwent Contrast Enhanced Mammography
  Interventions: Device: Contrast Enhanced Mammography

INTERVENTIONS:
Device: Contrast Enhanced Mammography — Contrast Enhanced Mammography

SUMMARY:
The study's objective is to compare the diagnostic accuracy of the contrast-enhanced mammography (CEM) , considering as reference the classification obtained with Vacuum Assisted Breast Biopsy (VABB).

DETAILED DESCRIPTION:
Breast cancer is the most diagnosed cancer in women and is one of the leading causes of morbidity and death from malignancy.

Improvement in survival and quality of life of patients with breast malignancies depends on the ability of imaging to diagnose the neoplasm in its early stages.

The main focus of imaging applied to the study of the breast is to obtain a good balance between the number of false positives and false negatives in the prediction of malignancy: good diagnostic performance should be achieved in identifying even small and insidious neoplasms without requiring excessive examinations for benign findings.

The main diagnostic method of screening for breast malignancy still remains mammography also considering its quick execution and low cost: however as is well known the diagnostic performance of mammography is highly impaired, in patients with dense breasts. The reduced sensitivity of mammography in women with dense breasts can result in a significant underdiagnosis rate, failing to prevent death due to breast cancer in a non-negligible number of women. The sensitivity of mammography is reported in the literature as between 62-68% in dense breasts: such performance is far too low to ensure adequate support in the management of breast malignancy; supplemental screening should be recommended in women with dense breasts.

For this purpose, a diagnostic technique called contrast-enhanced mammography (CEM) has been developed in recent years: CEM is based on the use of an iodinated contrast medium to assess the vascularity of any breast lesions and its first use was approved in 2011 by the food and drug administration (FDA).

The diagnostic performance of CEM in detecting and predicting the malignancy of breast lesions has been evaluated in many studies that have shown very promising result: CEM seems to provide excellent performance, particularly where conventional diagnostic methods seem to be struggling: the low sensitivity of mammography in dense breasts; the high operator dependence of breast ultrasound; the high cost, the high number of false positives and the time required to perform Magnetic Resonance Imaging (MRI).

The purpose of this studt is to assess the diagnostic performance of recombined CEM image, in predicting malignancy of breast lesions in a population mainly represented by patients with dense breasts.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast lesions, who underwent bilateral CEM
* Histological assessment

Exclusion Criteria:

* The subject is known to have risks of adverse effects with iodine contrast agents
* The subject has breasts too large to be adequately positioned on Full field digital mammography (FFDM) digital receptor without anatomical cut off during an FFDM examination

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of negative predictive value (NPV) of the CEM | 1 month
  Assessment of diagnostic accuracy of CEM in dense breasts considering as reference the classification obtained with VABB. Negative predictive value will be expressed as the proportion of patients classified as having no evidence of disease or Ductal Carcinoma In Situ (DCIS) at surgery among all patients with absence of contrast uptake at CEM

SECONDARY OUTCOMES:
Evaluation of sensitivity of CEM | 1 month
  Sensitivity will be expressed as the proportion of patients classified as positive with CEM, among all patients with malignant tumors classified with VABB (true positives)
Evaluation of specificity of CEM | 1 month
  Specificity will be expressed as the proportion of patients classified as negative with CEM, among all patients with benign tumors classified with VABB (true negatives)
Positive Predictive Value (PPV) of CEM | 1 month
  The positive predictive value will be expressed as the proportion of patients with malignant tumors classified with VABB among all patients classified as positive with CEM

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Cassano, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- Breast Imaging Division, Radiology Department, IEO European Institute of Oncology IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: No